CLINICAL TRIAL: NCT03682328
Title: Comparetive Study Between Vertebroplasty and Kyphoplasty in the Management of Osteoporotic Vertebral Body Fractures.
Brief Title: Vertebroplasty and Kyphoplasty in Osteoporotic Vertebral Body Fractures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud M. Gamal, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vertebroplasty and kyphoplasty
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Osteoporotic Fracture of Vertebra
Keywords: Vertebroplasty; Kyphoplasty; Osteoporosis; Vertebral fractures
MeSH Terms: conditions — Osteoporosis; Spinal Fractures | interventions — Vertebroplasty

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vertebroplasty (Active Comparator): Patients will be managed by equipment of vertebroplasty (Osteofix from Tsunami Medical Made in Italy which is composed of a packet of PMMA and ampule of MMA).
  Interventions: Procedure: vertebroplasty
- kyphoplasty (Active Comparator): Patients will be managed by equipment of kyphoplasty (Osteofix from Tsunami Medical Made in Italy which is composed of a packet of PMMA and ampule of MMA).
  Interventions: Procedure: kyphoplaty

INTERVENTIONS:
Procedure: vertebroplasty — Cement augmentation of the vertebral body
  Arms: vertebroplasty
Procedure: kyphoplaty — Cement augmentation of the vertebral body
  Arms: kyphoplasty

SUMMARY:
Vertebral body fractures are a major health care problem in all countries with incidence 1.4%. They are a common cause of severe debilitating pain, with consequent deteriorated quality of life, physical function and psychosocial performance.

Surgery is indicated in patients with vertebral body fracture, and concurrent spinal instability or neurologic deficit. The cornerstone of management for vertebral body fractures without neurological impairment is medical therapy, which include analgesics, bed rest, orthoses and rehabilitation. In the majority of patients such treatment modalities are effective. However, conservative management measures are not indicated for every type of fracture. For example, in older patients with vertebral fractures and cardio-respiratory disease it is not possible to prescribe bedrest for long period. Moreover, sometimes anti-inflammatory drugs are poorly tolerated by older patients, and bed rest can lead to further demineralization of the vertebrae, predisposing to future fractures.

Percutaneous minimally invasive vertebral augmentation methods for cement application into the vertebral body are a useful tool for the management of symptomatic fractures without neurological impairment when conventional measures of treatment can not be adopted. Two different percutaneous minimally invasive vertebral augmentation methods for cement application into the vertebral body for the management of symptomatic vertebral body fractures without neurological impairment have been developed, namely vertebroplasty and kyphoplasty.

Kyphoplasty and vertebroplasty have gained wide acceptance worldwide to manage patients without neurological impairment suffering from unmanageable pain caused by vertebral body fractures. Both procedures depend on mechanical stabilization of the fracture produced by cement injection into the fractured vertebral body.

Cement augmentation of the vertebral body by vertebroplasty and kyphoplasty was originally introduced for osteoporotic compression fractures, but surgeons have now applied these techniques as a method of enhancing anterior column support while avoiding the morbidity and complications associated with anterior approaches.

The mainstay of the controversy between kyphoplasty and vertebroplasty are height restoration, whether or not this height restoration is clinically significant, and the risks related to height restoration.

DETAILED DESCRIPTION:
This study is a Randomized interventional study to be done at neurosurgery department, Assiut Universitu Hospital, Assiut university, Egypt.

1. Vertebroplasty To achieve a low complication rate, the most important factor which influences the result of the vertebroplasty is the visualization of needle placement and cement application. Vertebroplasty may be performed using both fluoroscopy, and CT scanning to obtain an accurate visualization of needle position and cement distribution. The monitoring of the distribution of the cement under direct fluoroscopic control is another crucial aspect of the procedure, independently from the technique used for needle placement.

   Vertebroplasty can be performed under local anaesthesia or a combination of conscious sedation in most patients, and is therefore particularly useful in patients with risk factors for general anaesthesia. General anaesthesia is required only in patients unable to cooperate due to pain or in very agitated patients.

   The access path depends on the level of the vertebral segment to be injected. In the lumbar spine, a transpedicular route is preferred. In the thoracic vertebrae, an intercostovertebral access is recommended. In the cervical vertebrae, an anterolateral approach is used.

   The cement should be injected while in its tooth-paste like phase to minimize complications from extravasation in the surrounding tissues, as the flow characteristics of the cement change over the time.

   Cement injection may be stopped when the anterior two thirds of the vertebral body are filled and the cement is homogenously distributed between both endplates. During cement injection, continuous fluoroscopic monitoring is performed to immediately detect extravasations of cement. In case of extravasation, the procedure must be interrupted.

   A direct correlation between the risk of extraosseous extravasation and the amount of cement injection has been proposed, but, to date, no studies have addressed the specific issue of the volume of cement needed during vertebroplasty. Normally, 2.5-4 mL of cement should provide good filling of the vertebra and achieve both consolidation and pain relief in patients with osteoporotic fractures.
2. Kyphoplasty Kyphoplasty is normally performed under general anaesthesia in some patients as proper placement of the balloons is mandatory, and several steps need to be taken before cement can be injected.

A mono- or bilateral trans- or para-pedicular approach is used to insert a working cannula into the posterior aspect of the vertebral body. The procedure is performed under fluoroscopy or CT scan control. With reaming tools, two working channels within the anterior aspect of the vertebral body are produced, and the appropriate balloon is inserted. To reduce the fractured vertebra and to produce a cavity, the balloon is inflated using visual volume and pressure controls. The behaviour of the vertebral body is monitored under fluoroscopic control. Inflation is stopped when a pressure above 250 psi is obtained, when the balloon contacts the cortical surface of the vertebral body, or if the balloon expands beyond the border of the vertebral body, and if the height of the vertebra is restored. Successively, the balloons are retracted and cement polymethylmetacrylate (PMMA) is injected using a blunt cannula under continuous fluoroscopic control.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 60 years.
2. Sex: both males and females.
3. Compressive and burst vertebral body fractures without any neurological deficit.
4. Failure of medical treatment for at least 3-4 weeks

Exclusion Criteria:

1. Unmanageable bleeding disorder.
2. Improvement of the symptoms of the patient with conservative management.
3. Asymptomatic vertebral body fracture or presence of neurological deficit.
4. Local or generalized infection.
5. Known allergy to bone cement.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
back pain | up to 6 months
  Measuring and comparing the post-operative back pain via Visual analogue scales system

SECONDARY OUTCOMES:
kyphotic deformity | up to 6 months
  Measuring and comparing the post-operative via kyphotic deformity Cobb's angle.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla, MD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lieberman IH, Togawa D, Kayanja MM. Vertebroplasty and kyphoplasty: filler materials. Spine J. 2005 Nov-Dec;5(6 Suppl):305S-316S. doi: 10.1016/j.spinee.2005.02.020. PMID 16291128
- [Background] Phillips FM. Minimally invasive treatments of osteoporotic vertebral compression fractures. Spine (Phila Pa 1976). 2003 Aug 1;28(15 Suppl):S45-53. doi: 10.1097/01.BRS.0000076898.37566.32. PMID 12897474